CLINICAL TRIAL: NCT01909219
Title: A Randomized Controlled Trial Comparing Efficacy and Acceptability of Split and Standard Dose Sodium Picosulphate/Magnesium Citrate for Bowel Cleansing Prior to Colonoscopy: the MAGIC-P Multicenter Study
Brief Title: PMC Split Preparation for Colon Cleansing
Acronym: MAGIC-P
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Luigi Sacco University Hospital (Other)
Responsible Party: Principal Investigator, Gianpiero Manes, Medical Doctor, Luigi Sacco University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMC split
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Colon Cleansing
Keywords: preparation, cleansing, colon
MeSH Terms: interventions — picosulfate sodium; magnesium citrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: standard regimen (Active Comparator): Patients in the group A (standard regimen) will be instructed to take the two sachets of sodium picosulphate/magnesium citrate diluted in a glass of water 2-4 hours apart, starting at 5 pm the day before colonoscopy.
  Interventions: Drug: Sodium picosulphate/magnesium Citrate
- Group B (Active Comparator): Patients in the group B (split regimen) will be instructed to take the first sachet of sodium picosulphate/magnesium citrate at 7 pm the day before colonoscopy and the second one at 6 am in the morning on the day of colonoscopy.
  Interventions: Drug: Sodium picosulphate/magnesium Citrate

INTERVENTIONS:
Drug: Sodium picosulphate/magnesium Citrate — Comparison of two different dosing regimens of sodium picosulphate/magnesium citrate
  Other Names: Citrafleet

SUMMARY:
This is an endoscopist-blinded, prospective, multicenter study involving adult outpatients aiming at evaluating whether sodium picosulphate/magnesium citrate split dosing is associated to higher efficacy and acceptability in comparison to the standard dose regimen in bowel cleansing before colonoscopy

DETAILED DESCRIPTION:
Picosulphate/magnesium citrate is a very effective, safe and tolerated low-volume preparation for colon cleansing. This study evaluates whether split dosing is associated to a further increase in efficacy and acceptability in comparison to the standard dose regimen. This is a multicenter, randomized, single-blind study performed in 15 endoscopic services in Italy.

Adult outpatients undergoing colonoscopy will receive picosulphate/magnesium citrate either in the standard dosing (group A, two sachets the day before endoscopy), or in the split dosing (group B, the second dose in the morning of colonoscopy). Bowel cleansing will be assessed using the Boston Scale (BBPS) and rated as adequate if >2 in each segment. Patient acceptance, satisfaction, and related symptoms will be also recorded.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatients
* aged 18-85 yr
* undergoing elective colonoscopy

Exclusion Criteria:

* previous colon resection,
* ileus,
* intestinal obstruction,
* toxic megacolon,
* severe heart failure (NYHA Class III or IV),
* acute cardiovascular disease,
* uncontrolled arterial hypertension (systolic pressure >170 mmHg, diastolic pressure >100 mmHg),
* severe liver cirrhosis (Child-Pugh score C),
* renal failure (creatinine clearance<30 mL/minute),
* ascites,
* phenylketonuria,
* glucose-6-phosphate dehydrogenase deficiency,
* pregnant or breastfeeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Rate of adequate colon cleansing | 24 hrs
  The primary endpoint of the study was the quality of overall colon cleansing, assessed by the endoscopist. Colon cleansing quality was dichotomized as "adequate" (score > 2 in each colon segment) or "inadequate" (score < 2 in one or more colon segments

SECONDARY OUTCOMES:
Patients' acceptance, tolerability and compliance to the cleansing regimen | 24 hrs
  The overall tolerance of the preparation and the severity of symptoms during the preparation period will be rated on a scale ranging from 0 (no discomfort) to 3 (severe discomfort). Patient acceptance of the preparation will be evaluated by a questionnaire with a 5-point scale ranging from 1 (worse) to 5 (best), assessing interference with daily activity, palatability, easiness in taking the product and the adjunctive clear fluid, and taste of product. Moreover, a nurse will ask the patient whether s/he have completed the prescribed regimen: compliance will be defined as poor for patients who consume less than 75% of product. Willingness to repeat the same preparation in the future will be also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiero Manes, MD, Principal Investigator — Sacco Huniversity Hospital
Locations (2):
- Italy (2):
  - Luigi Sacco University Hospital, Milan, Milano
  - Luigi Sacco University Hospital, Milan

REFERENCES:
- [Derived] Manes G, Repici A, Hassan C; MAGIC-P study group. Randomized controlled trial comparing efficacy and acceptability of split- and standard-dose sodium picosulfate plus magnesium citrate for bowel cleansing prior to colonoscopy. Endoscopy. 2014 Aug;46(8):662-9. doi: 10.1055/s-0034-1365800. Epub 2014 Jul 14. PMID 25019969